CLINICAL TRIAL: NCT07329101
Title: Clinical Study to Evaluate the Safety, Pharmacokinetics and Efficacy of VC005 in Adolescent Subjects With Mild to Moderate Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC005-106
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VC005 (Experimental)
  Interventions: Drug: VC005

INTERVENTIONS:
Drug: VC005 — VC005 with Local topical application

SUMMARY:
This is a single arm, and open-label phase I study

ELIGIBILITY:
Inclusion Criteria:

* When giving informed consent, the age range is 12-18 years old (including 12 years old), with no gender restrictions;
* The subjects and their guardians voluntarily sign an informed consent form (dated), indicating that the subjects have been informed of all relevant parts of the study;
* All women and all men with the potential to conceive must be willing to use at least one highly effective method of contraception from the time of signing the informed consent form until 3 months after the last administration of the investigational drug

Exclusion Criteria:

* Subjects suspected to be allergic to VC005 gel or to excipients in VC005 gel, or with ≥ 2 kinds of drug allergy history in the past;
* The researchers believe that there may be skin injuries or abnormalities in the subjects that could affect the evaluation of the administration site of the investigational drug；
* The researchers believe that the subjects have clinically relevant skin diseases that are contraindicated in the study or affect the evaluation of the administration site, including but not limited to psoriasis, acne, dysplastic nevi, and skin cancer;

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC） | Day1，Day28
Peak Plasma Concentration (Cmax） | Day1，Day28

CONTACTS AND LOCATIONS:
Overall Officials: Liming Wu, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China